CLINICAL TRIAL: NCT03733769
Title: A Novel Approach for Transmuscular Quadratus Lumborum Block for Peri-operative Analgesia in Hip Surgery
Brief Title: A Novel Approach for Transmuscular Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmad Samir Alabd, assistant lecturer of anaesthesiology, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQL block in hip surgery
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Transmuscular Quadratus Lumborum Block Hip Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQL group (Experimental): transmuscular quadratus lumborum block as an alternative to lumbar plexus block for peri-operative analgesia in hip Surgery
  Interventions: Procedure: transmuscular quadratus lumborum block

INTERVENTIONS:
Procedure: transmuscular quadratus lumborum block — transmuscular quadratus lumborum block as an alternative to lumbar plexus block for peri-operative analgesia in hip Surgery

SUMMARY:
a novel approach for TQL (anterior Q.L) block aiming mainly for terminal branches of lumbar plexus. The technique is described as Para-Spinous Saggital Shift Q.L block, done at L4 transverse process level in saggital orientation.

DETAILED DESCRIPTION:
With this approach, we think it has advantages of easy identification, better caudal LA spread till under fascia iliaca, with the psoas major muscle provides a better protective barrier against accidental needle entry into the peritoneal cavity, the endpoint is injection within a fascial plane, rather than a specific motor response contact where the lumbar plexus stimulation is not sought, so there is minimal risk of nerve injury, inadvertent dural cuff puncture and intrathecal spread of local anesthetic. And finally optimal insertion of catheter in long axis of Q.L and psoas major if continuous analgesia is planned.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic patients, American Society of Anesthesiologists (ASA) physical status I-III, scheduled to undergo unilateral hip surgery.

Exclusion Criteria:

* History of neurological/neuromuscular, psychiatric disease, dementia preventing proper comprehension.
* Patients with Body Mass Index (BMI) <18.5 or >30 kg/m2.
* Coagulation disturbances (INR>1.4, platelet count<100 000).
* History of opioid dependence (opioid use within the last 4 weeks).
* History of allergies to study medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
peri-operative analgesia in hip Surgery | one month
  post-operative VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Emad A Abdelmonem, Study Chair — Alexandria faculty of medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Adhikary SD, Short AJ, El-Boghdadly K, Abdelmalak MJ, Chin KJ. Transmuscular quadratus lumborum versus lumbar plexus block for total hip arthroplasty: A retrospective propensity score matched cohort study. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):372-378. doi: 10.4103/joacp.JOACP_335_17. PMID 30386022
- [Background] Adhikary SD, El-Boghdadly K, Nasralah Z, Sarwani N, Nixon AM, Chin KJ. A radiologic and anatomic assessment of injectate spread following transmuscular quadratus lumborum block in cadavers. Anaesthesia. 2017 Jan;72(1):73-79. doi: 10.1111/anae.13647. Epub 2016 Oct 12. PMID 27730633
- [Background] Carline L, McLeod GA, Lamb C. A cadaver study comparing spread of dye and nerve involvement after three different quadratus lumborum blocks. Br J Anaesth. 2016 Sep;117(3):387-94. doi: 10.1093/bja/aew224. PMID 27543534